CLINICAL TRIAL: NCT06041893
Title: Haploidentical Hematopoietic Stem Cell Transplantation With Early Antithymocyte Globulin and Low Dose Post-transplant Cyclophosphamide
Brief Title: Haploidentical Hematopoietic Stem Cell Transplantation With Early ATG and Low Dose Post-transplant Cyclophosphamide
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KeonHee Yoo, Professor, Samsung Medical Center
Other Study IDs: SMC 2023-03-094-002
Record Dates: First submitted 2023-07-06; First posted 2023-09-18 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Haploidentical Hematopoietic Stem Cell Transplantation
Keywords: post transplant cyclophosphamide; antithymocyte globulin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — To confirm the recovery of immune function, T (including Treg, Tmemory), B, and NK cell counts will be checked before hematopoietic stem cell transplantation and 1, 3, 6, and 12 months after transplantation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ATG/LD-PTCy group: Patients undergoing haploidentical hematopoietic stem cell transplantation with ATG and low-dose post-transplant cyclophosphamide conditioning at the department of pediatrics, Samsung Medical Center
  Interventions: Drug: ATG-LDPTCy

INTERVENTIONS:
Drug: ATG-LDPTCy — antithymocyte globulin with low dose post-transplant cyclophosphamide

SUMMARY:
Aim of this study is to investigate the effect of early administration of anti-thymocyte globulin and post-transplant low-dose cyclophosphamide in heploidentical hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation from a haploidentical donor (haplo-HCT) are increasingly used in patients lacking a matched donor, but the optimal strategy needs to be defined. This study aims to investigate the outcome of haplo-HCT with early antithymocyte globulin and low dose posttransplant cyclophosphamide (ATG/LD-PTCy) in a single center.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing haploidentical hematopoietic stem cell transplantation with ATG and low-dose post-transplant cyclophosphamide conditioning at the department of pediatrics, Samsung Medical Center.

Exclusion Criteria:

* A clinical trial subject (legal representative, if applicable) who do not consent or is unable to give written consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing haploidentical hematopoietic stem cell transplantation with ATG and low-dose post-transplant cyclophosphamide conditioning at the department of pediatrics, Samsung Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2025-07-05 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Emgraftment Rate | From the date of transplantation until 28 days after transplantation
  cumulative incidence of donor-dominant engraftment by day 28 (by case)
Time to Engraftment | From the date of transplantation until first neutrophil count over 500/uL for 3 consecutive tays
  median time to neutrophil engraftment
Acute Graft-Versus-Host Disease | From the date of transplantation until 365 days after transplantation
  Incidence of acute GVHD ≥ grade 2
Chronic Graft-Versus-Host Disease | From the date of transplantation until the date of documentation of highest level of chronic GVHD, assessed up to 2 years after transplantation
  Incidence of moderate to severe chronic GVHD

SECONDARY OUTCOMES:
Rate of CMV infection | From the date of transplantation until 365 days after transplantation
  Rate of CMV infection
Rate of Hemorrhagic Cystitis | From the date of transplantation until 365 days after transplantation
  Rate of Hemorrhagic Cystitis

OTHER OUTCOMES:
Immune reconstitution | From the date of transplantation until 365 days after transplantation
  B cell, T cell (CD3+, CD4+, CD8+, Regulatory, Memory) NK cell count (of peripheral blood) at 1, 3, 6, 12 months post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Keon Hee Yoo, Professor, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided